CLINICAL TRIAL: NCT00992862
Title: A Relative Bioavailability Study of Moexipril HCl 15mg Tablets Under Fasting Conditions
Brief Title: A Relative Bioavailability Study of Moexipril HCl 15 mg Tablets Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Paddock Laboratories, Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: B035302
Record Dates: First submitted 2009-10-07; First posted 2009-10-09 (Estimated); Last update posted 2013-09-26 (Estimated); Status verified 2009-10

CONDITIONS: Healthy
MeSH Terms: interventions — moexipril; Tablets

ARMS (2):
- Moexipril HCl 15mg Tablets (Experimental)
  Interventions: Drug: Moexipril HCl 15mg Tablets, Paddock Laboratories, Inc.
- Univasc® 15mg Tablets (Active Comparator)
  Interventions: Drug: Univasc® 15mg Tablets

INTERVENTIONS:
Drug: Moexipril HCl 15mg Tablets, Paddock Laboratories, Inc.
  Arms: Moexipril HCl 15mg Tablets
Drug: Univasc® 15mg Tablets
  Arms: Univasc® 15mg Tablets

SUMMARY:
The purpose of this study is to compare the relative bioavailability of Moexipril HCl 15mg tablets (by Paddock Laboratories, Inc.) with that of Univasc® 15mg tablets (by Schwarz Pharma) following a single oral dose (1 x 15mg tablet) in healthy, adult subjects under fasting conditions.

ELIGIBILITY:
Inclusion Criteria:

* Good health as determined by lack of clinically significant abnormalities in health assessment performed at screening

Exclusion Criteria:

* Positive test results for HIV or Hepatitis B or C
* History of allergy or sensitivity to Moexipril HCl or related drugs

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60

PRIMARY OUTCOMES:
Bioequivalence according to US FDA guidelines

CONTACTS AND LOCATIONS:
Overall Officials: Kennedy, M.D., Principal Investigator — Novum Pharmaceutical Research Services
Locations (1):
- Novum Pharmaceutical Research Services, Pittsburgh, Pennsylvania, United States